CLINICAL TRIAL: NCT04901377
Title: A Prospective Multicenter Non-interventional Study to Evaluate User Satisfaction With Estradiol Valerate/ Dienogest in Real Clinical Practice to be Conducted in Russia
Brief Title: A Study to Gather Information About User Satisfaction in Women in Russia Who Take Estradiol Valerate/Dienogest
Acronym: Q-SWAN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21768
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Oral Contraception
MeSH Terms: interventions — estradiol valerate-dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined oral contraception: Estradiol valerate / Dienogest: Young women (18-35 years of age) using estradiol valerate / dienogest in real clinical practice.
  Interventions: Combination Product: Estradiol valerate/ Dienogest

INTERVENTIONS:
Combination Product: Estradiol valerate/ Dienogest — Combined hormonal contraceptive (combined oral contraceptives, COCs)
  Other Names: Qlaira®

SUMMARY:
Researchers want to learn more about user satisfaction in women in Russia who take estradiol valerate/ dienogest as a contraceptive in real conditions.

Estradiol valerate/ dienogest is a form of birth control. This is also known as a combined oral contraceptive (COC). Earlier studies showed that estradiol valerate/ dienogest has high level of protection from unplanned pregnancy. It is available for doctors to prescribe to women who want to take an oral contraceptive.

Estradiol valerate/ dienogest as a combined oral contraceptive (COC), works by stopping a process called ovulation. This is the process by which the ovaries release an egg. COCs are commonly used by young women to prevent pregnancy.

The researchers in this study will collect information from young women (18-35 years of age) in Russia who will start taking estradiol valerate/ dienogest.

The main purpose of this study is to find out about the women's satisfaction with taking estradiol valerate/ dienogest. To do this, the researchers will ask "how satisfied are you with the birth control method used during the study?". They will ask this question after the women have taken estradiol valerate/ dienogest for 3 and 6 months. The women willanswer this question using a rating scale ranging from 1 to 5, with 1 meaning "very dissatisfied" and 5 meaning "very satisfied".

This study will include young women (18-35 years of age) who want to use oral contraceptives and have been prescribed estradiol valerate/ dienogest by their doctor. None of the women in the study will have taken estradiol valerate/ dienogest within 1 month of joining the study.

In this study, it is expected that each woman will visit her study site 3 times. Each woman will be in the study for up to 6 months. All of the women will take estradiol valerate/ dienogest as prescribed by their doctors. There will be no other required procedures or treatments in this study which is not be used in usual practice.

During the study, the women will answer a question about how satisfied they are with estradiol valerate/ dienogest. They will also respond to some questionnaires. These will include a questionnaire about their menstrual bleeding patterns, sexual function. The doctors will:

* ask the women about any medical conditions they may have and what other contraceptives they took before they joined the study
* check the women's blood pressure and pulse rate
* ask a question about woman's intention to continue to use estradiol valerate/ dienogest and the reasons for discontinuation of estradiol valerate/ dienogest if it has happened

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 35 y.o.
* Indications for administration of estradiol valerate/ dienogest for the purpose of oral contraception.
* Patients who did not take estradiol valerate/ dienogest for at least one month before enrollment into the study.
* Signed informed consent to participate in the study

Exclusion criteria

* Participation in an investigational program with interventions outside of routine clinical practice.
* Contraindications to estradiol valerate/ dienogest according to the local market authorization.
* Any medical and non-medical reasons that according to the physician's judgment may prevent patient's participation in the non-interventional study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women 18 to 35 years of age who elect to use oral contraceptives will be enrolled after the decision for administration of estradiol valerate/ dienogest has been made by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
User satisfaction rates | up to 6 months
  User satisfaction rates assessed by subjects using an overall satisfaction rating (5-point Likert item) with the following question: "How satisfied are you with the birth control method used during the study?" Answers include: 1 - very dissatisfied; 2 - dissatisfied; 3 - neither satisfied nor dissatisfied; 4 - satisfied; 5 - very satisfied.
  Subjects selecting answers #4 or #5 (i.e., subjects expressing satisfaction) will count toward the overall satisfaction rate.

SECONDARY OUTCOMES:
Satisfaction rates assessed by physicians | up to 6 months
  Satisfaction rates assessed by physicians using an overall satisfaction rating (5-point Likert item) with the following question: "How satisfied are you with the birth control method used during the study?" Answers include: 1 - very dissatisfied; 2 - dissatisfied; 3 - neither satisfied nor dissatisfied; 4 - satisfied; 5 - very satisfied.
  Physicians selecting answers #4 or #5 (i.e., physicians expressing satisfaction) will count toward the overall satisfaction rate.
Bleeding profile | up to 6 months
  The bleeding profile during the previous 3 months and during therapy (visits 2,3), self-reported: regularity (regular, periodically absent, permanently absent); maximum bleeding duration (1-2 days, 3-5 days, 6-7 days, 8 days and more); maximum bleeding intensity (spotting, light bleeding, normal bleeding, heavy bleeding); painful bleeding (yes/ no); inter-menstrual bleeding (yes/ no).
Sexual function using FSFI | up to 6 months
  Sexual function using "Female Sexual Function Index" (FSFI).
Sexual function using ASQ | up to 6 months
  Sexual function using Atrophy Symptom Questionnaire (ASQ): dryness; sensitivity; irritation; dyspareunia; vaginal discharge (each symptom will be assessed with the following scale: 0 - normal, 1 - mild, 2 - moderate, 3 - severe).
Reasons for discontinuation | up to 6 months
Patient's intentions to continue to take estradiol valerate/ dienogest | up to 6 months
  yes / no

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here for access to information about Bayer's transparency standards and Bayer studies — https://clinicaltrials.bayer.com